CLINICAL TRIAL: NCT00304538
Title: A Phase 1b, Single-Blind Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of Three Separate Dose Levels of Very Low Dose-Glucagon Administered Subcutaneously Overnight for 6, 9 or 12 Hours in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Study of the Safety, Tolerability, Pharmacokinetics and Pharmacodynamic Activity of Very Low Dose-Glucagon in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: DiObex (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DIO-103
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2006-08-23 (Estimated); Status verified 2006-08

CONDITIONS: Type 1 Diabetes
Keywords: diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Glucagon

INTERVENTIONS:
Drug: very low dose (VLD) glucagon

SUMMARY:
The purpose of this study is to identify the safest dose of very low dose glucagon to prevent hypoglycemia in patients with Type I diabetes who use insulin pumps and to measure the the amount of glucagon in the blood and see how the body responds to the glucagon.

DETAILED DESCRIPTION:
Glucagon is currently used to treat severe hypoglycemia. DiObex believes that glucagon replacement therapy with very low doses of glucagon may prevent hypoglycemia without compromising effective glycemic control by insulin. In this study very low doses of glucagon will administered to Type I diabetics who use insulin pumps. The glucagon will be administered subcutaneously overnight for 6, 9 or 12 hours to see if the number of mild or impending hypoglycemia events can be safely decreased. Three different doses of glucagon will be compared to a control infusion.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, 18 to 55 years of age, requiring daily insulin for the management of type 1 diabetes mellitus for >10 years
2. On a stable basal insulin regimen using CSII therapy ("stable" defined as total daily dose of insulin not changed by more than ± 20% for 2 months prior to screening)
3. Glycosylated hemoglobin (HbA1c) ≤8.0%
4. Total daily insulin requirement of ≤1 unit/kg of body weight
5. Fasting C-peptide level of <1.0 ng/mL (<330 pmol/L) (may be done at screening or may be taken from subject's medical record if performed within the past 12 months)
6. Body mass index (BMI) ≤25.5 kg/m2 and body weight over past 6 months within ± 5%
7. Hemoglobin, hematocrit, and platelets within normal limits; no clinically significant abnormality of white blood cells (WBC) or differential
8. Serum chemistry results within normal limits except for liver enzymes [aspartate transaminase (AST) and alanine transaminase (ALT)] which must be within 2.5 times upper limit of normal (ULN) and creatinine which must be <1.6 mg/dL
9. Normal thyroid stimulating hormone
10. No history of HIV infection and negative results for hepatitis B and C
11. Negative serum pregnancy test, non-lactating, and using adequate contraception, if female and of child bearing potential (intact uterus and pre-menopausal)
12. Medications for the treatment of high blood pressure and/or dyslipidemia are allowed if regimen stable for 2 months prior to screening
13. Medically stable as determined by history and physical examination, including vital signs
14. Electrocardiogram (ECG) shows no acute ischemia or clinically significant abnormality
15. Willing and able to give written informed consent

Exclusion Criteria:

1. Participation in a clinical trial with or use of an investigational agent within 30 days of Study Visit 1.
2. History of atherosclerosis including coronary artery disease, angina pectoris, myocardial infarction, cerebrovascular accident, or transient ischemic attacks
3. History or symptoms of pheochromocytoma
4. History of any malignancy within 3 years except for basal cell skin cancer
5. Active infection, drug or alcohol abuse, eating disorder, or psychiatric disorder
6. Concomitant medications: systemic or potent topical steroids or medications that may affect blood glucose, e.g., sulfonylureas, alpha-glucosidase inhibitors, biguanides, meglitinides, thiazolidinediones
7. Any condition which increases the risk of participation in the trial in the opinion of the investigator -

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10
Dates: Start 2006-03; Study Completion 2006-07

PRIMARY OUTCOMES:
1) Evaluate the safety and tolerability of VLD-glucagon in doses of 2, 4 and 8 ng/kg/minute when infused overnight 2) Evaluate the PK profile in plasma of VLD-glucagon 3) Evaluate the pharmacodynamic activity of these doses by measuring glucose levels

SECONDARY OUTCOMES:
Compare the number of times and amount of time subjects have glucose levels < 70 mg/dL when treated with VLD-glucagon vs. the control infusion

CONTACTS AND LOCATIONS:
Overall Officials: Steven Edelman, MD, Principal Investigator — University of California, San Diego
Locations (1):
- University Of California, San Diego, San Diego, California, United States